CLINICAL TRIAL: NCT05245019
Title: Effects of Cardamom and Fennel on Salivary pH and Anti Microbial Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Dr Rabia Arshad, Associate Professor and Head, Department of Pharmacology, Altamash Institute of Dental Medicines. Karachi, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AIDM
Record Dates: First submitted 2022-01-25; First posted 2022-02-17 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Electrolyte Disturbance; Saliva Altered
MeSH Terms: interventions — Foeniculum vulgare fruit

STUDY DESIGN:
Intervention Model Description: Males & Females Patients ≥ 18 years Individuals not undergoing topical fluoride therapy, other chemotherapeutic procedures, antibiotics, and drugs having an effect upon the salivary function or salivary pH Individuals not suffering from any systemic diseases/ taking any medication that affects salivary secretion
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cardamom group (Experimental): the pH of saliva will be checked first then they r required to chew cardamom nd after 15 minutes again pH will be checked
  Interventions: Biological: cardamom
- fennel group (Experimental): the pH of saliva will be checked first then they r required to chew fennel and after 15 minutes again pH will be checked
  Interventions: Biological: fennel

INTERVENTIONS:
Biological: cardamom — cardamom is used as a flavoring agent in foods as well as for treating various cardiovascular, gastrointestinal, and neural problems
  Other Names: Elettaria cardamomum
  Arms: cardamom group
Biological: fennel — fennel is Known for its anti-inflammatory, anti-spasmodic, and analgesic properties, it is also widely used for treating gastroenteritis and indigestion.
  Other Names: Foeniculum vulgare
  Arms: fennel group

SUMMARY:
Dental caries is the most prevalent infectious disease related to oral health.. Although significant advances have been made on a global front to prevent caries, studies show its incidence is on the rise making it one of the major chronic diseases affecting all age groups. It possesses not only a great load concerning cost on developed nations but an increasing burden on developing nations. It largely affects children and the lower socioeconomic group hence demanding feasible and inexpensive ways to counter this growing ailment.

Dental caries is a multifactorial disease involving the interaction of the host, agent, and the environment. The primary etiologic agent implicated in dental caries is the streptococcus mutans and non-streptococcus species like Lactobacillus, Actinomyces, and Veillonella species. These oral microbes break down carbohydrates content in the diet, producing acids as by-products. The acids produced lower the pH of plaque and saliva resulting in the demineralization of enamel and dentine, finally enhancing the formation of cavities or dental caries.

The role of saliva in maintaining oral health has been studied extensively over time. The buffering capacity of saliva prevents the teeth from demineralization by maintaining the pH of the oral cavity thereby reducing the risk of dental caries. Since ancient times, medicinal plants and herbs have been used for maintaining oral health. Recent studies have shown fennel seeds and cardamom to play a significant role in regulating the pH of saliva and plaque, and ultimately preventing dental caries.

Cardamom (Elettaria cardamomum) is used as a flavoring agent in foods as well as for treating various cardiovascular, gastrointestinal, and neural problems. In addition, its extracts have shown antimicrobial activity against the principal pathogens causing dental caries and oral candidiasis. The commonest are S. mutans and Lactobacillus.

Fennel (Foeniculum vulgare) is a dry seed used in treating various ailments. Known for its anti-inflammatory, anti-spasmodic, and analgesic properties, it is also widely used for treating gastroenteritis and indigestion. Over time, it has been used in many oral care products for its antiseptic properties and as a breath freshener on its own. Studies have found fennel to not only inhibit the activity of streptococcus Mutans but also cause a significant rise in salivary pH hence depicting the anti-cariogenic activity.

Given the above literature, this study has been designed to record the effects of cardamom and fennel on the salivary pH and their anti-microbial activity on selected microbial species in our population.

DETAILED DESCRIPTION:
This study has been designed to evaluate the effects of cardamom and fennel on oral pH and microbes of the oral cavity.

OBJECTIVES OF THE STUDY:

1. To compare the change in pH of the saliva before and after Cardamom use
2. To compare the change in pH of the saliva before and after Fennel use
3. To compare the pH changes after fennel and cardamom use on patients' saliva
4. To evaluate the effects of Cardamom extract on oral pathogens (S. mutans and Lactobacillus)
5. To evaluate the effects of Fennel extract on oral pathogens
6. To compare the effects of Cardamom and Fennel extract on oral pathogens.

STUDY DESIGN:

Randomized clinical trial

INCLUSION CRITERIA:

1. Completely dentate individuals
2. Males & Females Patients ≥ 18 years
3. Individuals not undergoing topical fluoride therapy, other chemotherapeutic procedures, antibiotics, and drugs affecting the salivary function or salivary pH
4. Individuals not suffering from any systemic diseases/ taking any medication that affects salivary secretion (14).

METHODOLOGY:

Patients coming to the dental setting for a dental checkup or dental procedures, after written informed consent will be enrolled in the study. They will be requested not to take anything orally except plain water for an hour. After an hour they will be required to give salivary samples as control first (control salivary samples). pH will be measured of provided salivary samples with a portable digital pH meter.

Afterward, divided randomly into groups A with a minimum of 25 patients will be given Cardamom (one pod). The second group, Group B will be given Fennel (half teaspoon full, 1.3 grams) to be chewed for 10 minutes under the supervision of the researcher. The saliva will again be collected in clean containers and pH will be assessed.

For the second part of the study, the extract will be prepared with ten grams of fruit powder to be kept in 70% methanol (100ml) for 3 days, followed by filtration and proper storage. Bacteria will be grown from control salivary samples on the required agars. With micro-pathological techniques and expertise, the extract will be applied to the agar and the zone of inhibition will be measured in millimeters on inoculated agar plates with the agar well diffusion method. Standard strains as control will be taken from DDRL Lab. For positive control, Tablet Ciprofloxacin will be used. (12).

Data collected will be evaluated statistically using SPSS 26. For numerical values, mean with standard deviation, and for categorical values percentages will be calculated. To compare before and after paired T-test and to compare between the two treatments, students' T-test will be applied. A value equal to and greater than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Completely dentate individuals
2. Males & Females Patients ≥ 18 years
3. Individuals not undergoing topical fluoride therapy, other chemotherapeutic procedures, antibiotics, and drugs having an effect upon the salivary function or salivary pH
4. Individuals not suffering from any systemic diseases/ taking any medication that affects the salivary secretion

Exclusion Criteria:

1. Patients suffering from systemic diseases
2. Patients taking drugs that can effect ph. of saliva
3. Patients less then18 years of age -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
salivary pH | 1 Month
  Change in pH will be observed before and after cardamom and fennel chewing

SECONDARY OUTCOMES:
anti-microbial activity | 1 Month
  Anti-microbial activity of common oral pathogens will be assessed in vitro. The prepared extract will be applied on oral bacteria (Streptococcus mutans and Lactobacillus) grown on agar plates. After incubation, the zone of inhibition will be measured in millimeters with a measuring scale on inoculated agar plates with the agar well diffusion method. the collected measurements will be assessed for a maximum zone of inhibition in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: RABIA ARSHAD, Ph.D, Principal Investigator — ALTAMASH INSTITUTE OF DENTAL MEDICINE, KARACHI
Locations (1):
- Altamash Institute of Dental Medicine, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manohar R, Ganesh A, Abbyramy N, Abinaya R, Balaji SK, Priya SB. The effect of fennel seeds on pH of saliva - A clinical study. Indian J Dent Res. 2020 Nov-Dec;31(6):921-923. doi: 10.4103/ijdr.IJDR_185_19. PMID 33753665